CLINICAL TRIAL: NCT07090174
Title: A Single-Arm, Open-Label Clinical Phase II Trial of the Safety and Immunogenicity of PDS0101 in People Living With HIV
Brief Title: Testing for Safety and Immune Effects of PDS0101, an Anti-HPV Therapy, Among People Living With HIV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of Puerto Rico (Other); Montefiore Medical Center (Other); Albert Einstein College of Medicine (Other); University of California, San Diego (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); National Cancer Institute (NCI) (NIH); Emory University (Other); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-08027893; U54CA242639 (NIH); ULACNet-203 (Other: National Cancer Institute)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: HPV Associated Cancers; HIV (Human Immunodeficiency Virus); Anal Cancer; Cervical Cancer; HPV 16 Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anus Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PDS0101 HPV 16 immunotherapeutic agent (Experimental)
  Interventions: Biological: PDS0101

INTERVENTIONS:
Biological: PDS0101 — PDS0101 is an HPV 16-targeted immunotherapy administered as two subcutaneous injections of 0.5 mL each (total 1.0 mL). Each dose contains 3.0 mg of Versamune®, a proprietary cationic lipid nanoparticle adjuvant, and 2.7 mg of HPVmix, a blend of HPV16 E6 and E7 proteins. Versamune® enhances antigen uptake and dendritic cell activation, promoting T-cell priming and memory formation. In preclinical studies, subcutaneous administration resulted in low systemic bioavailability (<6%) and efficient dendritic cell uptake, consistent with a favorable safety profile. PDS0101 has been studied in a completed Phase I trial in HIV-uninfected women with high-risk HPV and cervical intraepithelial neoplasia (CIN) I. Each participant in this study will receive three doses, spaced 21 days apart (± 7 days) unless there has been Grade 3 or greater toxicity at least possibly related to the study agent.
  Other Names: Versamune® + HPVmix

SUMMARY:
This study is testing the immunotherapeutic agent, PDS0101, in adults living with HIV who are also infected with human papillomavirus (HPV) type 16. The purpose of the study is to learn whether PDS0101 is safe and whether it can help the body's immune system respond to HPV 16. Researchers will enroll 27 adults between the ages of 25 and 65 who have been receiving antiretroviral therapy (ART) for at least 12 months, have a cluster of differentiation 4 (CD4) cell count of at least 200 cells/mm³, and have an HIV viral load below 200 copies/mL. All participants must have HPV 16 detected in the cervix, vagina, or anus. Some participants will have high-grade squamous intraepithelial lesions (HSIL), a condition that can lead to cancer. At least 10 participants will have cervical HSIL, and at least 10 will have anal HSIL. Participants with both cervical and anal HSIL will count in both groups. Others may have HPV 16 without HSIL.

This is a single-arm, open-label trial, which means that all participants will receive the same treatment, and both the investigators and the participants will know what the treatment is. Each participant will receive three doses of the PDS0101 vaccine. Participants who receive at least one dose will be included in the study's main safety analysis. If a participant does not receive all three doses and does not experience a serious side effect related to the vaccine (defined as a Grade 3 or higher toxicity), that participant may be replaced to make sure that 27 participants either complete the full vaccination schedule or experience a primary safety event. Participants who do have a qualifying safety event will not be replaced. Even if someone stops the study early, their data will still be included in the final analysis.

The main goals of this study are to evaluate the safety of PDS0101 and to measure the immune response it produces. The safety evaluation includes monitoring for serious or unexpected side effects, especially those that are Grade 3 or higher in severity. The immune response will be assessed by looking at how the body's T cells respond to HPV 16 after PDS0101 administration. The total time a participant is involved in the study includes the PDS0101 administration period and several follow-up visits, which may take place over the course of several months. This research may help inform future strategies for preventing or treating HPV-related disease in people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* HPV 16 detected on anal swab, cervical swab or vaginal swab ≤90 days of registration. (Note: HPV 16 detected on this swab can be from the screening evaluation or through standard of care assessments. The HPV 16 assay must be FDA-cleared and report HPV 16 results separately. The assay must be performed in a CLIA-certified laboratory.)
* Cervical HSIL cohort: CIN III/carcinoma in situ (CIS), CIN II/III, or CIN II with positive p16 stain diagnosed on cervical biopsy ≤90 days of registration and detection of cervical or vaginal HPV 16.
* Cervical HSIL cohort: HSIL must occupy <50% circumference of the cervical squamocolumnar junction, and adequate colposcopy with visualization of the endocervical HSIL margins. (Note: Participants with cervical HSIL occupying ≥50% of the circumference of cervical squamocolumnar junction and/or inadequate visualization of the endocervical HSIL margins are not eligible for this protocol.)
* Anal HSIL cohort: anal intraepithelial neoplasia (AIN) III, AIN II/III, or AIN II with positive p16 stain diagnosed on anal or perianal biopsy ≤90 days of registration and detection of anal HPV 16.
* Anal HSIL cohort: HSIL must occupy <50% circumference of the squamocolumnar junction. (Note: Participants with anal HSIL occupying ≥50% of the circumference of cervical squamocolumnar junction are not eligible for this protocol.)
* Ages 25-65 years (i.e., no longer eligible on the 66th birthday).
* HIV infection with receipt of antiretroviral therapy for at least 12 months.
* CD4+ T-cell count ≥200 cells/mm3 ≤45 days of registration.
* Plasma HIV-1 RNA <200 copies/mL ≤45 days of registration.
* Participants must meet the following laboratory parameters ≤45 days before enrollment:

  1. Absolute neutrophil count: ≥1,500/mm3
  2. Platelets: ≥100,000/mm3
  3. Hemoglobin >12.5 g/dL for men and >11.5 g/dL for women
  4. Estimated glomerular filtration rate (eGFR) >70 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation or serum creatinine <1.2 x upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) (SGOT), and alanine aminotransferase (ALT) (SGPT), <1.5 x ULN
  6. Total bilirubin <1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (or Karnofsky ≥70%).
* Willingness to comply with three-dose immunotherapeutic agent schedule and subsequent study visits.
* The effects of PDS0101 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception prior to study entry and for at least 120 days after the last dose of study treatment. Women of childbearing potential must have a negative urine pregnancy test (β-human chorionic gonadotropin) within 24 hours prior to registration and prior to visits on Days 1, 22, 43, 57, and 127. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately and will not receive any additional doses of immunotherapeutic agent. Women who become pregnant and partners of male participants who become pregnant will be followed to assess pregnancy outcomes.
* Ability to understand and the willingness to sign a written informed consent form (ICF).

Exclusion Criteria:

* AIDS-defining condition within 6 months prior to study entry.
* Receipt of blood products within 6 months of enrollment or are currently taking immune suppressants.
* History of HPV-related cancer or suspected cancer of the cervix, anus, vagina, vulva, penis, or oropharynx.
* Current diagnosis of cancer or prior invasive cancer > T1 stage (other than non-melanoma skin cancer) that has required active treatment within the past 3 years.
* Suspicion of invasive cancer of the cervix, vulva, vagina, perianus or anal canal. (Note: Concomitant vulvar, vaginal, or perianal HSIL is not exclusionary.)
* Surgical or ablative treatment for anal or cervical HSIL within 180 days of study entry.
* Prior receipt of any doses of a licensed or experimental HPV immunotherapeutic agent. (Note: Prior receipt of licensed prophylactic HPV vaccines is permitted.)
* Planned use of intravaginal, vulvar, perianal or intra-anal imiquimod or 5-fluorouracil or another topical therapeutic agent with possible activity against HPV disease, or their use within ≤90 days of entry.
* Receipt of a live vaccine within 30 days prior to the first dose of treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Coordination and timing of COVID-19 vaccination should be based on local Investigator clinical assessment and judgment.
* Received immunotherapy/immunomodulatory or immunosuppressive agents (e.g., IFNs, tumor necrosis factor, interleukins, immunoglobulins or other biological response modifiers [GM-CSF, granulocyte-macrophage colony-stimulating factor]) within 6 weeks prior to administration of the first study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 30 days prior to the first dose of study treatment. (Note: Participants who entered the follow-up phase of an investigational study may participate as long as it has been 30 days after the last dose of the previous investigational agent.)
* Is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Current or recent use of intra-articular, topical, or inhaled corticosteroids is acceptable.
* Participants known to be positive for Hepatitis B antigen (HBsAg)/Hepatitis B virus (HBV) DNA or active Hepatitis C. Active Hepatitis C (HCV) is defined by a known positive HCV antibody result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
* Plan to relocate during study period.
* Acute medical conditions that would require exclusion from participation based on the opinion of the supervising physician.
* Potential participants receiving any other investigational agents may be excluded in the opinion of the supervising physician.
* Use of opioids within 2 weeks prior to enrollment. (Note: Medically assisted therapy for opioid use disorder or alcohol use disorder (e.g., stable methadone or buprenorphine/naloxone) are not exclusionary. The rationale for excluding other opioid use is to allow appropriate grading of injection-related pain.)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Current bacterial sexually transmitted infection (STI) requiring treatment (participants may participate after adequate treatment, at the discretion of the treating provider).
* Pregnant or breastfeeding, unwilling/unable to use contraception, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of any study treatment.

  a) For the purpose of this study, a WOCBP (i.e., fertile) is defined as the period following menarche and until becoming post-menopausal unless permanently sterile. Acceptable methods of birth control for this study include: i) Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

ii) A post-menopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the post-menopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

iii) Use of a barrier (diaphragm or condom) with spermicide iv) Combined hormonal (estrogen and progestogen) contraception associated with inhibition of ovulation v) An intrauterine device/system vi. An oral, transdermal, or injectable contraceptive vii. A vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success.

b) For the purpose of this study, a man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy.

i. Male participants must agree to use a condom as an effective method of contraception throughout the study and for at least 120 days after the last dose of study treatment.

* Use of anticoagulants other than non-steroidal anti-inflammatory drugs or aspirin.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of Grade 3 or greater adverse events (AE) at least possibly related to PDS0101. | 127 days
  Adverse events will be scored according to CTCAE v5.0 grading (Grade 1-Mild, Grade 2-Moderate, Grade 3-Severe, Grade 4-Life-threatening, and Grade 5-Fatal) except for injection site reactions (ISRs) grading, wherein they will be reviewed against 2007 FDA guidance. Skin discoloration is common with PDS0101, therefore skin discoloration (ISRs including erythema or pigment changes) >10 cm and induration >10 cm will not count as a primary safety endpoint. However, all of the detailed AEs will be reported as a supporting analysis including all ISRs. For the primary safety analysis, we will include all participants who receive at least one dose of PDS0101. Participants who only receive 1-2 doses who discontinue PDS0101/study participation for reasons other than a primary safety event will be replaced to assure 27 participants who receive all 3 doses or discontinue PDS0101 after 1-2 doses because of a primary safety event; those with primary safety event after 1-2 doses won't be replaced.
Tolerability: Proportion of participants who receive all three doses. | 127 days
  Participants who do not receive the first dose will be excluded from all analyses.

SECONDARY OUTCOMES:
Proportion of participants with an immunotherapeutic agent-induced response. | 127 days
  Immunotherapeutic agent-induced response is defined as a ≥ 3-fold increase over baseline at ≥ 1 of the 4 post-dose administration visits by either interferon gamma (IFN-γ) or granzyme ELISPOT assays, with background subtracted. The proportion with a response by each assay will be reported separately and at each post-study immunotherapeutic agent administration visit.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Ellsworth, MD, MS, Principal Investigator — Weill Medical College of Cornell University; Timothy Wilkin, MD, MPH, Study Chair — University of California, San Diego
Locations (3):
- United States (2):
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be shared 3 months after we have published on the specific aims of the study through the duration of the NIH award (U54242639).
Access Criteria: Researchers granted access to the data will be required to use it solely for research purposes, ensuring that no individual participants are identifiable. They must also implement appropriate security measures, such as using password-protected servers and files, to safeguard the data. Upon completion of the analyses, the data must be returned or destroyed. Released datasets will be subject to stringent safeguards to ensure compliance with the Health Insurance Portability and Accountability Act (HIPAA). Additionally, a data-sharing agreement will be required, specifying that the data is used exclusively for research purposes and that no participants are identifiable. A data management plan will also be necessary to ensure the continued security and confidentiality of the data, as well as to outline the process for returning or destroying the data once the analysis is complete.